CLINICAL TRIAL: NCT07344389
Title: The Effect of Virtual Reality Application on Body Composition, Functional Capacity, Balance, and Participation in Children With Hyperlipidemia
Brief Title: Virtual Reality Intervention in Children With Hyperlipidemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Duygu Korkem, Assistant Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-424
Record Dates: First submitted 2025-12-26; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hyperlipidemia in Children
Keywords: Hyperlipidemia; Virtual Reality Training; Pediatric Rehabilitation; Physical Activity; Participation
MeSH Terms: conditions — Hyperlipidemias; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Virtual Reality Training Group (Experimental): Participants allocated to the experimental group will receive a virtual reality-based exercise program in addition to continuing their usual dietary regimen. The intervention will be delivered for 8 weeks, twice per week, with each session lasting 40 minutes. Virtual reality training will be provided using an interactive system designed to promote physical activity through game-based exercises. All assessments will be conducted by a blinded assessor.
  Interventions: Other: Virtual Reality Training
- Control Group: Conventional Physiotherapy Home Exercise Group (Active Comparator): Participants allocated to the control group will continue their usual dietary regimen and will receive general conventional physiotherapy exercises designed for home practice. These exercises will be demonstrated to the participants and their families at baseline. No virtual reality training will be provided to this group. All assessments will be conducted by a blinded assessor.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Virtual Reality Training — The intervention consists of an 8-week virtual reality-based exercise program using the Microsoft Kinect system for children with hyperlipidemia. Sessions will be conducted twice per week, each lasting 40 minutes. The Kinect system will track participants' three-dimensional body movements in real time using an infrared depth sensor and RGB camera. Game-based activities will be projected onto a wall, and participants will perform exercises by interacting with virtual tasks such as boat navigation and ball games. The system will provide real-time visual feedback to reinforce correct movements and correct improper movement patterns. The program is designed to promote physical activity, improve motor skills, and support cardiovascular fitness in an engaging and enjoyable environment.
  Arms: Experimental Group: Virtual Reality Training Group
Other: Conventional Physiotherapy — Participants in the control group will continue their usual dietary regimen and receive a conventional physiotherapy home exercise program. The program will consist of general exercises aimed at maintaining physical activity and functional capacity and will be demonstrated to the participants and their caregivers at baseline. No virtual reality-based intervention will be provided during the study period. Participants will be encouraged to perform the exercises at home throughout the 8-week study duration.
  Arms: Control Group: Conventional Physiotherapy Home Exercise Group

SUMMARY:
Children with hyperlipidemia have elevated blood lipid levels, which increase the risk of developing cardiovascular diseases later in life. Since the atherosclerotic process begins in childhood, early identification and effective management of risk factors such as physical inactivity are essential. Regular physical activity has been shown to improve lipid profiles, reduce cardiovascular risk, and support healthy body composition in children. However, long-term lifestyle and medical treatments may reduce motivation and participation, especially in pediatric populations.

Virtual reality-based exercise programs provide an engaging and interactive environment that can increase motivation and active participation in rehabilitation. Virtual reality applications allow children to perform functional movements through game-based activities while receiving visual and auditory feedback, which may enhance motor learning, balance, and functional capacity. These applications are widely used in pediatric rehabilitation and have the potential to improve adherence to exercise programs.

Participation in daily life activities at home, school, and in the community is an important component of child development. According to the International Classification of Functioning, Disability and Health (ICF), participation refers to involvement in life situations. Children with chronic health conditions may experience limitations in participation due to physical, environmental, or motivational factors. However, participation levels of children with hyperlipidemia have not been sufficiently investigated.

The purpose of this study is to investigate the effects of a virtual reality-based exercise program on body composition, functional capacity, balance, and participation in children with hyperlipidemia. The findings of this study may contribute to the development of effective, enjoyable, and sustainable rehabilitation approaches for improving physical health and participation in daily life activities in this population.

DETAILED DESCRIPTION:
Hyperlipidemia in childhood is an increasingly prevalent metabolic disorder associated with early initiation of the atherosclerotic process and an elevated risk of cardiovascular disease in adulthood. Since atherosclerosis begins in childhood, early identification and management of hyperlipidemia, particularly through lifestyle-based interventions, are critical for long-term cardiovascular health. Regular physical activity is known to positively influence lipid metabolism by reducing triglyceride levels, increasing high-density lipoprotein cholesterol, and improving endothelial function. However, adherence to long-term exercise and lifestyle recommendations in children is often limited due to low motivation and sedentary behaviors.

Virtual reality-based exercise interventions offer an innovative and engaging approach to increase physical activity participation in children. By providing immersive, interactive, and gamified environments, virtual reality applications can enhance motivation, enjoyment, and adherence to exercise programs. Virtual reality training integrates core principles of motor learning, including task repetition, goal-oriented movement, multisensory feedback, and active participation, which are essential for improving physical function and promoting sustained behavioral change.

This prospective randomized controlled study is designed to investigate the effects of an 8-week virtual reality-based exercise program on physical and functional outcomes in children with hyperlipidemia. Participants will be randomly allocated to either a virtual reality training group or a control group using computer-based randomization software. All assessments will be conducted by an assessor blinded to group allocation. To minimize confounding effects related to nutrition, participants in both groups will continue their usual dietary management throughout the study period.

The intervention group will participate in virtual reality-based exercise sessions twice weekly for eight weeks, with each session lasting approximately 40 minutes. Training will be delivered using the Microsoft Kinect system, a markerless motion capture technology capable of detecting and analyzing three-dimensional body movements in real time. The system enables participants to interact with virtual environments through whole-body movements and provides immediate visual and auditory feedback. Exercise sessions will include a variety of game-based activities that promote aerobic exercise, dynamic balance, coordination, and functional movement patterns. The intensity and content of the sessions are designed to support cardiovascular fitness while maintaining engagement and enjoyment.

Outcome assessments will be performed at baseline, immediately after the 8-week intervention period, and at an 8-week follow-up to examine both short-term and sustained effects of the intervention. The study evaluates changes in body composition, physical activity level, functional capacity, balance, speed and agility, flexibility, body image perception, and participation across home, school, and community settings, in accordance with the International Classification of Functioning, Disability and Health (ICF) framework.

Participation is a key component of child development and health, encompassing involvement in daily life situations and social roles. Children with chronic health conditions often experience reduced participation, influenced by both personal and environmental factors. Despite the growing prevalence of pediatric hyperlipidemia, participation patterns and environmental influences in this population have not been adequately explored. This study aims to address this gap by examining participation outcomes alongside physical and functional measures.

By integrating virtual reality-based exercise into the management of pediatric hyperlipidemia, this study seeks to determine whether an engaging, technology-assisted intervention can improve physical health parameters while also supporting participation and functional involvement in daily life. The findings may contribute to the development of innovative, child-centered rehabilitation and preventive strategies for managing hyperlipidemia and reducing long-term cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8-14
* Diagnosed with hyperlipidemia
* No condition preventing physical activity in the past seven days
* Children and families who volunteer to participate in the study will be included.

Exclusion Criteria:

* Children with any physical, neurological, or cognitive illness
* Children who do not wish to participate in the study
* Children who do not complete the assessment will be excluded

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Body Weight | 8 week
  Body weight will be measured using the Tanita body composition analyzer (MC-780MA) and recorded in kilograms.
Physical activity | 8 week
  Children's physical activity levels will be assessed using the Physical Activity Questionnaire for Children (PAQ-C). The PAQ-C is a self-report instrument designed to evaluate general physical activity levels in children and adolescents over the previous 7 days. It consists of 10 items, of which 9 are used to calculate the activity score. The first item includes a culturally adapted activity checklist consisting of 14 common activities and is scored on a 5-point scale (1 = no activity, 5 = 7 times or more). The remaining 8 items assess physical activity during specific periods of the day or week, such as physical education classes, recess, after school, evenings, and weekends, and are also rated on a 5-point scale. The final PAQ-C score is calculated as the mean of items 1-9, with higher scores indicating higher levels of physical activity.
Functional capacity | 8 week
  Functional capacity will be assessed using the Six-Minute Walk Test (6MWT). The 6MWT is a simple, practical, and objective exercise test widely used to evaluate functional exercise capacity in children. Participants will be instructed to wear comfortable clothing and appropriate footwear. They will rest before the test, and heart rate, blood pressure, oxygen saturation (SpO₂), and perceived dyspnea using the Modified Borg Scale will be recorded before and after the test. Participants will be asked to walk back and forth along a marked 30-meter flat corridor for six minutes, aiming to cover the longest possible distance. Standardized verbal encouragement will be provided at each minute. The total distance walked in six minutes will be recorded in meters.
Participation | 8 week
  Participation and environmental factors will be assessed using the Participation and Environment Measure for Children and Youth (PEM-CY). The PEM-CY is a parent-reported questionnaire designed to evaluate participation of children and adolescents aged 5-17 years in home, school, and community settings, as well as environmental influences on participation. The participation section includes 10 activities for the home setting, 5 for the school setting, and 10 for the community setting. For each activity, parents report the frequency of participation over the past four months, the child's level of involvement using a five-point Likert scale, and whether they desire a change in the child's participation. The PEM-CY has demonstrated acceptable validity and reliability in Turkish populations.
Body Mass Index (BMI) | 8 week
  Body mass index will be calculated as body weight divided by height squared (kg/m²) using measurements obtained from the Tanita body composition analyzer (MC-780MA).
Body Fat Composition | 8 week
  Body fat composition will be assessed using the Tanita body composition analyzer (MC-780MA). Measurements will include total body fat percentage (%) and total body fat mass (kg), which together will be used to evaluate changes in overall adiposity.

SECONDARY OUTCOMES:
Body Image | 8 week
  Body image will be measured using the Children's Body Image Scale. There are separate versions of the scale for boys and girls. The scale contains 7 gender-specific images in anatomical position. There are 7 male and 7 female photos on the scale for each version. Each photo represents a different BMI range. The images are ranked from A to G according to increasing BMI.
Static Balance | 8 week
  Balance will be assessed using the Flamingo Balance Test. The test requires a wooden beam measuring 50 cm in length and 4 cm in height, and a stopwatch. Participants will be asked to stand barefoot on the beam for one minute, balancing on one leg while the other leg is flexed at the knee and held with the hand on the same side, mimicking a flamingo stance. Before the test, one practice trial will be provided to familiarize the child with the procedure. The test begins with a start command and is interrupted each time balance is lost, defined as the free leg touching the ground. After each loss of balance, the test is resumed until a total of one minute is completed. The score is recorded as the number of balance attempts within one minute. If balance is lost more than 15 times within 30 seconds or if the child falls, the test is terminated and a score of zero is recorded. The test is performed for both legs.
Dynamic balance | 8 week
  Dynamic balance will be assessed using the Y Balance Test. Participants will stand on one leg with both hands placed on their hips, positioning the great toe of the stance foot at the center starting line. While maintaining single-leg stance, participants will reach as far as possible with the free limb in the anterior, posteromedial, and posterolateral directions. The maximum reach distance in each direction will be measured with a measuring tape and recorded. The procedure will be repeated for the opposite lower extremity. Trials will be repeated if the participant fails to maintain balance, moves or lifts the stance foot, touches the ground with the reaching foot before reaching the maximum distance, or fails to return the reaching foot to the starting position. Lower extremity length will be measured from the anterior superior iliac spine to the medial malleolus for score normalization. The composite reach distance will be calculated as [(maximum anterior + maximum posteromedial +
Speed and agility | 8 week
  Speed and agility will be assessed using the Single-Leg Side Hop Test on the preferred leg. Participants will stand on their preferred leg with their hands placed on their hips, while the non-stance leg is held in neutral hip position with the knee flexed at 90 degrees. While maintaining this position, participants will be instructed to hop laterally to the right and left of a marked line as many times as possible within 15 seconds. A stopwatch will be used to time the test, and the number of correctly performed hops will be recorded. The test will be terminated if the participant removes their hands from their hips or if the stance foot loses its position or drops below the required level.
Flexibility | 8 week
  Flexibility will be assessed using the Sit-and-Reach Test. This test is commonly used to evaluate flexibility of the hamstring and posterior lower limb muscle groups. Participants will be barefoot and dressed in comfortable clothing, seated on the floor in a long-sitting position with the ankles positioned in neutral. They will be instructed to lean forward from the hips and reach as far as possible without bending the knees, holding the final position for approximately two seconds. The test will be performed twice, and the best distance reached will be recorded in centimeters.

IPD SHARING:
Plan to Share IPD: No